CLINICAL TRIAL: NCT05949918
Title: Efficacy of a Stage-Matched Intervention Based on The Transtheoretical Model of Change in Dietary Fat Reduction Among Female High School Students: A Randomized Controlled Trial
Brief Title: Efficacy of a Stage-Matched Intervention Based on The Transtheoretical Model of Change in Dietary Fat Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Mohammed Baqer Habeeb Abd Ali, Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: Dietary Fat Reduction
Record Dates: First submitted 2023-06-28; First posted 2023-07-18 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Dietary Fat Reduction

STUDY DESIGN:
Who Masked: Participant
Masking Description: The researchers will use two groups (study and control) in which participants will be randomly selected and assigned in each of the study and control groups using simple random sampling.
  The study intervention will be designed based on each Stage of Change of the Transtheoretical Model of Change in that participants in each Stage of Change will receive the intervention that matches the Stage of Change they would be in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Precontemplation, Contemplation, Preparation, Action, and Maintenance-based intervention (Experimental): The intervention that would consider the Processes of Change that people use when they would be in the Precontemplation Stage of Change.
  Interventions: Behavioral: Stage-matched interventions
- Contemplation-based intervention (Experimental): The intervention that would consider the Processes of Change that people use when they would be in the Contemplation Stage of Change.
  Interventions: Behavioral: Stage-matched interventions
- Preparation-based intervention (Experimental): The intervention that would consider the Processes of Change that people use when they would be in the Preparation Stage of Change.
  Interventions: Behavioral: Stage-matched interventions
- Action-based intervention (Experimental): The intervention that would consider the Processes of Change that people use when they would be in the Action Stage of Change.
  Interventions: Behavioral: Stage-matched interventions
- Maintenance-based intervention (Experimental): The intervention that would consider the Processes of Change that people use when they would be in the Maintenance Stage of Change.
  Interventions: Behavioral: Stage-matched interventions

INTERVENTIONS:
Behavioral: Stage-matched interventions — The study intervention will be designed based on each Stage of Change of the Transtheoretical Model of Change in that participants in each Stage of Change will receive the intervention that matches the Stage of Change they would be in.
  A 12-week interval would be considered between administering the intervention and posttest 1 and the same interval would be used between posttest 1 and posttest 2.

SUMMARY:
This study aims to examine the efficacy of a Stage-Matched Intervention based on The Transtheoretical Model of Change in dietary fat reduction among female high school students.

DETAILED DESCRIPTION:
This study aims to examine the efficacy of a Stage-Matched Intervention based on The Transtheoretical Model of Change in dietary fat reduction among female high school students.

The study intervention will be designed based on each Stage of Change of the Transtheoretical Model of Change in that participants in each Stage of Change will receive the intervention that matches the Stage of Change they would be in.

A 12-week interval would be considered between administering the intervention and posttest 1 and the same interval would be used between posttest 1 and posttest 2.

ELIGIBILITY:
Inclusion Criteria:

* High school male students who do not experience any psychiatric-mental disorder.

Exclusion Criteria:

* High school male students who experience any psychiatric-mental disorder.

Ages: 15 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — High school male students who do not experience any psychiatric-mental disorder.
Enrollment: 144 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-03-24 (Actual); Study Completion 2024-03-24 (Actual)

PRIMARY OUTCOMES:
Stages of Change Scale for Dietary Fat Reduction | 6 months
  Stages of Change Scale for Dietary Fat Reduction measures individuals' readiness to reduce dietary fat.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Baghdad, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided